CLINICAL TRIAL: NCT01060592
Title: Effect on Early Weight Loss by Adjusting Gastric Band During Surgery
Brief Title: LapBand Adjustment to Improve Early Weight Loss
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Crospon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-02
Record Dates: First submitted 2010-01-30; First posted 2010-02-02 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Gastric Band; LapBand; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stoma Adjustment at Surgery (Experimental): The first band adjustment will be made at surgery versus historical controls where the adjustment is not made for 3-4 weeks post-surgery. EndoFLIP device (FDA Device Listing Number : D091203)will be used to make the adjustment.
  Interventions: Device: EndoFLIP device (FDA Device Listing Number : D091203)
- Historic (No Intervention): Weight loss profile over time for 50 patients in the first 12 months after surgery as derived from historic control records. Band adjustments are made in a heuristic fashion during the year after surgery using the experience of surgeon alone

INTERVENTIONS:
Device: EndoFLIP device (FDA Device Listing Number : D091203) — The EndoFLIP balloon catheter will be introduced to the band and used to permit the band stoma size to be adjusted to 7mm.
  Arms: Stoma Adjustment at Surgery

SUMMARY:
Subjects having a gastric band fitted will have the first band adjustment done at surgery. The stoma will be set to 7mm using the EndoFLIP system to measure stoma size. Thereafter, band adjustments will be made using an adjustment chart, created at surgery, which shows stoma size versus band fill, to make adjustments in the normal follow-up visits. It is hypothesized that an early adjustment at surgery will promote earlier weight loss, and result in fewer band adjustments being required in the first year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing gastric band surgery
* Over 18 years of age

Exclusion Criteria:

* Actively bleeding varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Snow, DO FACOS, Principal Investigator — AIGB; John O'Dea, PhD, Study Director — Crospon
Locations (1):
- Specialty Surgery of Fort Worth, Hurst, Texas, United States

REFERENCES:
- [Result] Snow RG, O'Dea J. Does Intraoperative Gastric Band Adjustment to a Targeted Stoma Size Improve Weight Loss? One-year Results of a Feasibility Trial Bariatric Times. 2012;9(1):10-12.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 pts recruited between Oct 2009 and Jan 2010
Pre-assignment Details: N/A - Single arm non-randomized study
Groups:
- Stoma Adjustment at Surgery: The first band adjustment will be made at surgery versus historical controls where the adjustment is not made for 3-4 weeks post-surgery
- Historic: Weight loss profile over time for 50 patients in the first 12 months after surgery as derived from historic control records
Period: 4-6w
Arm/Group | Stoma Adjustment at Surgery | Historic
Started | 35 | 49
Completed | 23 | 39
Not Completed | 12 | 10
Period: 12m
Arm/Group | Stoma Adjustment at Surgery | Historic
Started | 35 (For some pts, %EWL were not taken/available in the 4-6w period but were available for the 12m period) | 49 (For some pts, %EWL were not taken/available in the 4-6w period but were available for the 12m period)
Completed | 35 | 31 (Historic data was not available at 12m for 18 of the historic controls)
Not Completed | 0 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Historic | Stoma Adjustment at Surgery | Total
Number analyzed (Participants) | 49 | 35 | 84
Age Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.6) | 40.1 (11.6) | 42.8 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 64
  Male | 13 | 7 | 20
Region of Enrollment [Number; unit: participants]
  United States | 49 | 35 | 84

OUTCOME MEASURES:

1. Primary Outcome: %Excess Weight Loss 4-6 Weeks After Surgery (Large and Small Bands)
Time Frame: 4-6 weeks post surgery
Measure: Mean (Standard Deviation); unit: %EWL
Arm/Group | Historic | Stoma Adjustment at Surgery
Number analyzed (Participants) | 39 | 23
%EWL | 15.63 (8.9) | 20.8 (10.8)

2. Secondary Outcome: Number of Band Adjustments Required in the First Year After Surgery
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Number of Adjustments
Arm/Group | Historic | Stoma Adjustment at Surgery
Number analyzed (Participants) | 49 | 35
Number of Adjustments | 6.47 (3.15) | 6.66 (2.9)

3. Primary Outcome: %Excess Weight Loss 4-6 Weeks After Surgery (Small Bands Only)
Time Frame: 4-6 weeks post surgery
Measure: Mean (Standard Deviation); unit: %EWL
Arm/Group | Historic | Stoma Adjustment at Surgery
Number analyzed (Participants) | 28 | 16
%EWL | 16.33 (9.54) | 23.07 (11.59)

4. Primary Outcome: % Excess Weight Loss 12 Months After Surgery (Large and Small Bands)
Time Frame: 12m post surgery
Measure: Mean (Standard Deviation); unit: %EWL
Arm/Group | Historic | Stoma Adjustment at Surgery
Number analyzed (Participants) | 31 | 35
%EWL | 48.3 (15) | 50.4 (24.5)

5. Primary Outcome: % Excess Weight Loss 12 Months After Surgery (Small Bands Only)
Time Frame: 12m post surgery
Measure: Mean (Standard Deviation); unit: %EWL
Arm/Group | Historic | Stoma Adjustment at Surgery
Number analyzed (Participants) | 26 | 23
%EWL | 48.71 (15.61) | 60.32 (22.77)

ADVERSE EVENTS:
Arm/Group | Historic | Stoma Adjustment at Surgery
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/35
Other Adverse Events (participants affected / at risk) | 0/49 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No